CLINICAL TRIAL: NCT02890875
Title: Efficacy and Safety of Ethanol Lock Therapy for the Prevention of Central Line-associated Bloodstream Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Berkeley Limketkai, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 38195
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Catheter-Related Infections
Keywords: ethanol lock; parenteral nutrition
MeSH Terms: conditions — Catheter-Related Infections; Hyperphagia | interventions — Vascular Access Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ethanol lock (Active Comparator): 70% ethanol
  Interventions: Other: Ethanol lock
- Heparin lock (Active Comparator): Heparinized saline (100 U/mL)
  Interventions: Other: Heparin lock

INTERVENTIONS:
Other: Ethanol lock
  Arms: Ethanol lock
Other: Heparin lock
  Arms: Heparin lock

SUMMARY:
Patients on long-term parenteral nutrition (PN) are at high risk for central line-associated bloodstream infections (CLABSI). This study evaluates the efficacy and safety of ethanol lock therapy for CLABSI prophylaxis in adult patients on PN.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (ages 18-80) on PN with silicone-based central venous catheters

Exclusion Criteria:

* Weight ≤ 50 kg
* Allergy/hypersensitivity/intolerance to ethanol or heparin
* Pregnancy or breastfeeding
* Patient taking metronidazole, disulfiram, or isoniazid
* History of alcohol abuse
* History of heparin-induced thrombocytopenia (HIT) or have an active hypocoagulable state

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Central line-associated bloodstream infection | 12 months

SECONDARY OUTCOMES:
Hospitalization | 12 months
SIRS/sepsis | 12 months
Catheter-related complication | 12 months
New self-reported symptoms | 12 months

OTHER OUTCOMES:
Microorganism (blood culture, if obtained for clinical reasons) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Berkeley Limketkai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States